CLINICAL TRIAL: NCT03240614
Title: PreOxygenation for Airway Management: High Flow Versus Conventional Preoxygenation Therapy
Brief Title: PreOxygenation for EndoTracheal Intubations
Acronym: POET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic and loss of funding
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: POET1
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2021-03

CONDITIONS: Intubation Complication; Preoxygenation; Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Will test preoxygenation using High Flow Nasal Cannulae, Non-rebreather mask and Bag-Valve-Mask
Who Masked: Outcomes Assessor
Masking Description: Interventions will be labeled using a Letter key so the analysis of the dataset by our statistician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- BMI <30 no lung disease (Active Comparator): Patients with a BMI <30 with no lung disease
  Interventions: Device: Non-rebreather oxygen mask; Device: Bag-valve-mask; Device: High Flow Nasal Cannulae
- BMI <30 with lung disease (Active Comparator): Patients with a BMI <30 with lung disease
  Interventions: Device: Non-rebreather oxygen mask; Device: Bag-valve-mask; Device: High Flow Nasal Cannulae
- BMI 30-35 with no lung disease (Active Comparator): Patients with a BMI between 30 and 35 with no lung disease
  Interventions: Device: Non-rebreather oxygen mask; Device: Bag-valve-mask; Device: High Flow Nasal Cannulae
- BMI 30-35 with lung disease (Active Comparator): Patients with a BMI between 30 and 35 with lung disease
  Interventions: Device: Non-rebreather oxygen mask; Device: Bag-valve-mask; Device: High Flow Nasal Cannulae
- BMI >35 with no lung disease (Active Comparator): Patients with a BMI> 35 with no lung disease
  Interventions: Device: Non-rebreather oxygen mask; Device: Bag-valve-mask; Device: High Flow Nasal Cannulae
- BMI >35 with lung disease (Active Comparator): Patients with a BMI> 35 with lung disease
  Interventions: Device: Non-rebreather oxygen mask; Device: Bag-valve-mask; Device: High Flow Nasal Cannulae

INTERVENTIONS:
Device: Non-rebreather oxygen mask — This intervention will be preoxygenation using a Non-rebreather that will be placed upon the participant for preoxygenation. The oxygen flow will be set at 60 L/min and the participant will be preoxygenated for a total of 3 minutes. After 3 minutes, an ABG will be taken and labeled as Intervention A.
Device: Bag-valve-mask — This intervention will be preoxygenation using a BVM apparatus for preoxygenation for 3 minutes. At the end of 3 minutes an ABG will be obtained.
Device: High Flow Nasal Cannulae — This intervention will be preoxygenation using High Flow Nasal Cannulaes at an FiO2 of 100%. The oxygen flow will be set at 60 L/min and the participant will be preoxygenated for a total of 3 minutes. After the 3 minutes, an ABG will be taken and labeled as Intervention C.

SUMMARY:
Hypoxemia is a life threatening complication during emergency airway management. Despite advances in technology and training, hypoxemia still occurs in up to a quarter of all intubations placing patients at high risk for damage to vital organs and death. A key method in the prevention of hypoxemia is known as preoxygenation which has been shown to decrease the incidence of hypoxemia. Currently there are two conventional methods for preoxygenation in the literature, however recently a new method has been described as a possible alternative method. What is unclear in the literature is if one modality is superior than the other for preoxygenation. The goal of this interventional study is to determine if one method of preoxygenation is superior to the other. This is a 3 arm interventional cross over designed study comparing three interventional methods for preoxygenation. Non-rebreather mask, bag-valve mask and high flow nasal cannulae.

DETAILED DESCRIPTION:
In emergency and critical care medicine, one of the most common incidences of severe hypoxemia occurs during the process of endotracheal intubations. Endotracheal intubations, also known as insertion of a breathing tube, is a life saving technique used in medicine to help maintain oxygen delivery, to protect lungs from injury, for patients to safely undergo anesthesia for surgeries, as well as to help rest critically ill patients to allow their bodies time to recover. Despite advances in the field of medicine, the process of placing a breathing tube in emergency situations is still associated with an increase risk of hypoxemia up to 26.7%. This places patients at significant risk for cardiac dysrhythmia, brain damage and hemodynamic decompensation which may ultimately result in death. A UK national review of emergency intubations identified hypoxemia as a cause of death in 50% of intensive care intubations and 27% of Emergency Department intubations. Therefore, it is imperative to improve and develop methods to minimize hypoxemia during airway management.

A vital component used to minimize the risk of hypoxemia during endotracheal intubations is preoxygenation. Preoxygenation is a method to to prolong the time to oxygen desaturation by replacing the lung volume with 100% oxygen compared to 21% oxygen (room air) through the administration of supplemental oxygen. This increases the reservoir of oxygen in the lungs that the body can use to prolong their time to desaturation. Studies have shown a good preoxygenation technique can increase the time to oxygen desaturation from 0.6 min to 8 min in a non obese patient. This remarkable impact at preventing hypoxemia has made preoxygenation the gold standard to minimize hypoxemia during airway management.

Historically preoxygenation with bag-valve-mask ventilation (BVM) and an oxygen non-rebreather mask has been the standard for preoxygenation. Recently, the use of high flow nasal cannulaes have been used for preoxygenation however it is unclear in the literature if one provides a superior preoxygenation compared to another. In an effort to determine the best preoxygenation modality for airway management, the investigators will conduct a 3 arm interventional crossover designed study to compare preoxygenation using a non-rebreather mask, BVM and HFNC in 150 patients. To determine which modality provides the best preoxygenation, arterial blood gases will be taken after each intervention and compared against each other.

Given the high propensity for hypoxemia during airway management in the obese and disease lung population, this protocol will have specific groups based on their BMI (<30, 30-35 and >35) as well as the presence of lung disease based upon their PaO2/FiO2 ratio (< 300 lung disease or >300 no lung disease).

However, due to the pandemic, we had to pause recruitment, a decision was made to do an power analysis with the number of patients we had recruited and a decision was made to collapse the study and report or findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pre-existing arterial line
* Age > 18
* Able to provide consent

Exclusion Criteria:

* Acute respiratory distress Defined as RR >30, Baseline oxygen requirements >50%, current use of High Flow Nasal Cannulae or Non-invasive ventilation for respiratory support
* Decreased level of consciousness GCS <13
* Possible exclusion if the allocation to prespecified groups are filled
* Contraindication for high oxygen therapy Severe Chronic Obstructive Pulmonary Disease with documented CO2 retention based on outpatient ABG History of Bleomycin use
* Significant hemodynamic instability Lactate > 3 mmol/L Norepinephrine dose >0.2 mcg/kg/min or equivalent dose of other vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
PaO2 | An ABG will be taken 3 min after preoxygenation in the NRB and HFNC group. The ABG will be taken once the ETO2 is >85% in the BVM group. Pooled data will be collected at the conclusion of the study to be analyzed within 6 months of completion.
  Partial pressure of arterial oxygen

SECONDARY OUTCOMES:
PaCO2 | An ABG will be taken 3 min after preoxygenation in the NRB and HFNC group. The ABG will be taken once the ETO2 is >85% in the BVM group. Pooled data will be collected at the conclusion of the study to be analyzed within 6 months of completion.
  Partial pressure of arterial carbon dioxide
Patient comfort | At the conclusion of all interventions the data will be collected on each individual participant. Pooled data will be collected at the conclusion of the study to be analyzed within 6 months of completion.
  Numeric scoring of patient comfort for each intervention

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gebremedhn EG, Mesele D, Aemero D, Alemu E. The incidence of oxygen desaturation during rapid sequence induction and intubation. World J Emerg Med. 2014;5(4):279-85. doi: 10.5847/wjem.j.issn.1920-8642.2014.04.007. PMID 25548602
- [Background] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Background] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948